CLINICAL TRIAL: NCT01040052
Title: A Bridging Study to Assess the Safety of the Vaccine Adacel® in a Clinical Trial
Brief Title: A Study to Assess the Safety of Adacel® Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TD532; U1111-1111-6093 (Other: WHO)
Record Dates: First submitted 2009-12-21; First posted 2009-12-25 (Estimated); Results first posted 2011-03-29 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Diphtheria; Tetanus; Pertussis
Keywords: Diphtheria; Tetanus; Pertussis; Adacel®
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — adacel; Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental)
  Interventions: Biological: Adacel® (Tetanus, Reduced Diphtheria Toxoid and Acellular Pertussis)

INTERVENTIONS:
Biological: Adacel® (Tetanus, Reduced Diphtheria Toxoid and Acellular Pertussis) — 0.5 mL, Intramuscular
  Other Names: Adacel®

SUMMARY:
The objective of this study is to describe the safety of Adacel® vaccination in adults subjects in Vietnam. This study is conducted in accordance with Vietnamese regulation in support to Adacel® registration.

Primary objective:

To monitor the adverse effects of the vaccine ADACEL® from day 0 to day 30 after immunization.

DETAILED DESCRIPTION:
Participants will receive a single dose of Adacel® vaccine and will be followed closely during 30 minutes post-vaccination period; a home visit will be made daily during 7 days following vaccination in order to monitor safety.

An additional visit will be conducted 30 days post-vaccination to collect safety information.

ELIGIBILITY:
Inclusion Criteria :

* Male or female (not pregnant) from 18-45 years of age.
* Healthy, with no current illnesses.
* Have not been immunized against diphtheria, pertussis and tetanus in the past 5 years.
* Women of childbearing age will agree to use birth control during the study.
* In good health, as verified by the following criteria: Heart rate, blood pressure, temperature and health history.
* Able to understand and comply with requirements of the study.
* A voluntary consent form is required before participating in the study.

Exclusion Criteria :

* History of allergy to any ingredient in the vaccine.
* A positive pregnancy test (for women of childbearing age) or women who are breastfeeding.
* Compromised immune system due to treatment of a progressive disease.
* Currently on oral or injected steroids, inhaled high-dosage steroids or other immunodeficiency or toxic drugs.
* History of taking Immunoglobulin or other products during the 3 months prior to participating in the study.
* Received other vaccines during the 4 months prior to participating in the study.
* Has an acute or chronic condition that affects safety (including but not limited to: chronic liver disease, some kidney pathologies, progressive or unstabilized nerve disorders, diabetes and organ transplants).
* Experienced a severe adverse event after receiving ADACEL® vaccine.
* History of acute illness with temperatures over 37.5ºC during the week before receiving the vaccine.
* Human immunodeficiency virus (HIV) infection.
* History of alcohol or drug addiction during the past 5 years.
* Plans to travel outside of the study area between shots and visits.
* History of Guillain-Barré syndrome.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Việt Trì, Phu Tho, Vietnam

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 06 to 13 December 2009 in 1 medical center in Vietnam.
Pre-assignment Details: A total of 30 participants who met the inclusion and exclusion criteria were enrolled, vaccinated, and evaluated.
Groups:
- ADACEL® Vaccine Group: All participants received a single dose of ADACEL® vaccine on Day 0.
Period: Overall Study
Arm/Group | ADACEL® Vaccine Group
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ADACEL® Vaccine Group
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.1 (5.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Region of Enrollment [Number; unit: participants]
  Vietnam | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting at Least One Solicited Local or Systemic Reaction Post-Vaccination With ADACEL® Vaccine
Description: Solicited injection site reactions: Pain, itchiness, erythema (redness), and swelling. Solicited systemic reactions: Headache, body ache and muscle weakness, tiredness, chill, nausea, vomiting, rash, itchiness, anorexia, sore and swollen joints, diarrhea, lymph node swelling, and fever (temperature).
Time Frame: Days 0-7 Post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | ADACEL® Vaccine Group
Number analyzed (Participants) | 30
Participants
  Any Solicited Injection Site Reaction | 27
  Any Injection Site Pain | 27
  Grade 3 Inj. site pain (hindered daily activities) | 0
  Any Itchiness | 1
  Grade 3 Itchiness (hindered daily activities) | 0
  Any Erythema | 1
  Grade 3 Erythema (hindered daily activities) | 0
  Any Swelling | 1
  Grade 3 Swelling (hindered daily activities) | 0
  Any Solicited Systemic Reaction | 5
  Any Headache | 2
  Grade 3 Headache (hindered daily activities) | 0
  Any Body Ache or Muscle Weakness | 1
  Grade 3 Body Ache or Muscle Weakness | 0
  Any Tiredness | 4
  Grade 3 Tiredness (hinders daily activities) | 0
  Any Chills | 1
  Grade 3 Chills (hinders daily activities) | 0
  Any Nausea | 0
  Grade 3 Nausea (hinders daily activities) | 0
  Any Vomiting | 0
  Grade 3 Vomiting (hinders daily activities) | 0
  Any Rash | 0
  Grade 3 Rash (hinders daily activities) | 0
  Any Itchiness | 0
  Grade 3 Itchiness (hinders daily activities) | 0
  Any Anorexia | 1
  Grade 3 Anorexia (hinders daily activities) | 0
  Any Sore and Swollen Joints | 0
  Gr 3 Sore and Swollen Joints (hinders activities) | 0
  Any Diarrhea | 0
  Grade 3 Diarrhea (hinders daily activities) | 0
  Any Lymph Node Swelling | 0
  Grade 3 Lymph Node Swelling (hinders activities) | 0
  Any Fever | 1
  Grade Fever (hinders daily activities) | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination up to 30 days post-vaccination.
Arm/Group | ADACEL® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 27/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADACEL® Vaccine Group (N=30)
Headache (Nervous system disorders) | 2 (2)
Tiredeness (General disorders) | 4 (4)
Injection site pain (General disorders) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications